CLINICAL TRIAL: NCT02992847
Title: Evaluation of Potential Accumulation of Gadolinium (Dotarem and Multihance) in the French Observatory of Multiple Sclerosis (Www.Ofsep.Org/)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0646
Record Dates: First submitted 2016-10-19; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Gadolinium based contrast agent; MRI; Dentate nucleus
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dotarem: At least 5 injection with Dotarem exclusively
  Interventions: Other: Unenhanced MRI
- Multihance: At least 5 injection with Multihance exclusively
  Interventions: Other: Unenhanced MRI

INTERVENTIONS:
Other: Unenhanced MRI

SUMMARY:
Several recent studies have shown an increase in the signal intensity of the unenhanced T1-weighted magnetic resonance images in the brain of patients with normal renal functions and a breakdown of the blood-brain barrier. This hyper-intensity was specifically related to an accumulation of gadolinium based contrast agent. These studies were mainly conducted in patients with primary or secondary brain tumor. Multiple sclerosis is a particular model since it involves patients with a break of the blood-brain barrier, a long life expectancy, and who received many injections of contrast enhancing agents. In this context, it appears fundamental to know whether contrast agents accumulate in the brain for this disease. The French Observatory of Multiple Sclerosis is particularly suited to test this hypothesis, with homogeneous MRI data over several centers in France, and optimized sequences of 3D-T1 without injection. The purpose of this study is to evaluate the accumulation of two commonly used gadolinium based contrast materials (Dotarem and Multihance) in patients with multiple sclerosis, who received at least 5 injection of exclusively one of these contrast material.

ELIGIBILITY:
* Inclusion Criteria:
* Clinical diagnosis of Multiple sclerosis
* At least 5 MR imaging with the same Gadolinium based contrast agent (either Dotarem or Multihance)
* Have performed an unenhanced T1-weighted image before Gadolinium based contrast agent injection according to the OFSEP protocol
* Exclusion Criteria:
* Never experienced other contrast agent then the one specified by the group to which they belong (either Dotarem, or Multihance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the French observatory of multiple sclerosis (www.ofsep.org/)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Mean signal intensity in the dentate nucleus, pons, globus pallidus, and thalamus on unenhanced T1-weighted images after unenhanced MRI (magnetic resonance imaging), (no measurement unit) | 12 months after last injection of contrast material for enhanced MR acquisition
  Operator defined region of interest measure of signal intensity on unenhanced T1-weighted images after MR acquisition

SECONDARY OUTCOMES:
EDSS (Expanded Disability Status Scale) score | 12 months after last injection of contrast material for enhanced MR acquisition